CLINICAL TRIAL: NCT04093011
Title: Perioperative Outcome of Congenital Heart Disease Surgery in Childhood: Results From a Chinese Cross-regional Cohort Study
Brief Title: Perioperative Outcome of Congenital Heart Disease Surgery in Childhood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator, Peking Union Medical College
Other Study IDs: TedaICH-Thousands of plans
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Congenital Heart Disease Surgery — Patients with congenital heart disease will undergo congenital heart disease surgery.

SUMMARY:
Congenital heart disease is the most common congenital malformation in the world with high morbidity and mortality. However, there is no data to assess the perioperative outcome of congenital heart disease surgery among Chinese cross-regional population. This study aims to investigate the perioperative outcome of congenital heart disease surgery in childhood from a chinese cross-regional cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subject was aged 1 week-18 years
* Subjects underwent congenital heart disease surgery;
* Available data to investigate perioperative outcome.

Exclusion Criteria:

* Cardiac reoperation;
* Emergency surgery;
* Interventional procedure within prior 30 days prior to surgery;
* Missing outcome data.

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients aged 1 week-18 years underwent congenital heart disease surgery from different Chinese regions.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of systemic inflammatory response syndrome | postoperative day 7 or hospital discharge, whichever occurred first.
  Systemic inflammatory response syndrome was determined mainly on (i) Core temperature of >38.5°C or <36°C measured by rectal, oral, or central catheter probe; (ii) Tachycardia, defined as a mean heart rate >2 SD above normal for age in the absence of external stimulus, chronic drugs, or painful stimuli; or otherwise unexplained persistent elevation over a 0.5- to 4-hr time period, or for children <1 yr old: bradycardia, defined as a mean heart rate <10th percentile for age in the absence of external vagal stimulus; or otherwise unexplained persistent depression over a 0.5-hr time period; (iii) Mean respiratory rate >2 SD above normal for age, the prolonged mechanical ventilation defined as ventilation duration > 48 hrs, or unplanned re-intubation for an acute process not related to underlying neuromuscular disease or the receipt of general anesthesia; (iv) Leukocyte count elevated or depressed for age or >10% immature neutrophils.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, MD, Study Director — Peking Union Medical College
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality, China